CLINICAL TRIAL: NCT05061784
Title: Revisiting the Evidence for Routine Transcervical Thymectomy for the Prevention of Thymic Carcinoid Tumours in MEN-1 Patients a Case Series
Brief Title: Routine Transcervical Thymectomy in MEN-1 Patients
Status: Completed | Type: Observational
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Rajeev Parameswaran, Assistant Professor and Head & Senior Consultant, National University Health System, Singapore
Other Study IDs: exempt from review
Record Dates: First submitted 2021-09-02; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Multiple Endocrine Neoplasia Type 1 (MEN-1); Thymic Carcinoid
Keywords: Routine transcervical thymectomy
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MEN-1 patients who underwent routine thymectomy during parathyroidecotmy: A case series was built after review of available literature by searching four databases (PubMed, Embase, Medline and Cochrane Library) for observational studies or case reports on routine prophylactic TCT for MEN-1 and the development of thymic carcinoids.
  Interventions: Procedure: Routine thymectomy, which has been performed

INTERVENTIONS:
Procedure: Routine thymectomy, which has been performed — There is no intervention

SUMMARY:
A case series was built after review of available literature by searching four databases (PubMed, Embase, Medline and Cochrane Library) for observational studies or case reports on routine prophylactic TCT for MEN-1 and the development of thymic carcinoids.

DETAILED DESCRIPTION:
Introduction and Importance Malignant thymic carcinoids are uncommon but important entities among patients with multiple endocrine neoplasia type 1 (MEN-1). Current treatment guidelines advise the performance of a routine transcervical thymectomy (TCT) during parathyroidectomy, to prevent its development, although data on the yield of this prophylactic TCT is scarce. We aimed to revisit available literature to investigate and summarize the efficacy of routine TCT during neck exploration for parathyroidectomy, for the prevention of thymic carcinoid tumours among MEN-1 patients.

Methods A case series was built after review of available literature by searching four databases (PubMed, Embase, Medline and Cochrane Library) for observational studies or case reports on routine prophylactic TCT for MEN-1 and the development of thymic carcinoids.

ELIGIBILITY:
Inclusion Criteria:

* Studies including MEN-1 patients who underwent a routine thymectomy during parathyoidectomy

  * We accepted randomized controlled trials or observational studies that included patients of any age who underwent a routine TCT in the setting for MEN-1, published as full-length articles in peer-reviewed journals, which mentioned data on thymic carcinoid tumours.

Exclusion Criteria:

* We excluded reviews, letters, conference proceedings and non-English publications.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We accepted randomized controlled trials or observational studies that included patients of any age who underwent a routine TCT in the setting for MEN-1, published as full-length articles in peer-reviewed journals, which mentioned data on thymic carcinoid tumours.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Incidence of thyme carcinoid | The timeframe will be from date of transcervical thymectomy until the date of documented diagnosis of diagnosis of thymic NET; progression of disease or date of death from any cause, whichever came first, assessed up to 100 months.
  Retrospective review of published studies

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
We will not be collecting data; just studies that have already been published